CLINICAL TRIAL: NCT03171714
Title: Derma-Stent Novel Abscess Packing Device (Pilot Study)
Brief Title: Derma-Stent Novel Abscess Packing Device
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aaron Brody, MD, MPH (Other)
Collaborators: Mar-Med (Unknown)
Responsible Party: Sponsor-Investigator, Aaron Brody, MD, MPH, Assistant Professor, Wayne State University
Organization: Wayne State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 091016M1F
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Cutaneous Abscess
Keywords: Drainage Catheter

STUDY DESIGN:
Intervention Model Description: Phase 1 - Pilot Trial:
  As this device has never been used on humans, the investigators will first deploy a pilot, uncontrolled trial of 10 subjects to assess for safety, and further refine outcome measures. The same protocol will be followed as the controlled trial, except the randomization.
  Phase 2 - Controlled Trial: 25 patients in each arm:
  1. Novel silicon packing device
  2. Usual Care, cotton gauze packing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Derma-Stent (Experimental): The novel silicon packing device made of a nonabsorbent material to pack a drained abscess for healing.
  Interventions: Device: Derma-Stent
- Usual Care, cotton gauze packing (Active Comparator): Standard of care to pack a drained abscess for healing.
  Interventions: Device: Usual care, cotton gauze packing

INTERVENTIONS:
Device: Derma-Stent — The novel device will facilitate self removal by patients, as it has a narrower profile, and, as a nonabsorbent material, will not become saturated with bodily fluids. Although it will not absorb body fluids
  Arms: Derma-Stent
Device: Usual care, cotton gauze packing — Standard gauze packing used to pack a drained abscess.
  Arms: Usual Care, cotton gauze packing

SUMMARY:
In this research study, a device called the Derma-Stent will be tested. The sponsor of the study, Mar-Med Company, will supply the device. This device is used to drain a cutaneous abscess, which is a skin infection that results in buildup of pus under the skin. Currently, the normal treatment for this abscess is to cut and drain and the wound, and later pack the wound with gauze. Packing is done to prevent the pus to accumulate again. But regular gauze is difficult for patient to remove themselves, so another visit to the doctor is usually necessary. The Derma-Stent device will be tested to see how easily patients can remove this by themselves and if it is less painful and more effective than normal gauze packing.

DETAILED DESCRIPTION:
Background:

Cutaneous abscess is an infectious condition that affects millions of people each year, and the incidence is on the rise. Between 1993 and 2005, the annual number of emergency department (ED) visits for skin and soft tissue infections increased from 1.2 to 3.4 million, and this largely attributed to a rise in the prevalence of Methicillin Resistant Staphylococcus Aureus (MRSA) in the community.

The standard treatment for cutaneous abscess is incision and drainage at bedside in the ED. Following this procedure, many clinicians insert a strip of gauze, known as packing, to maintain the open surgical incision, enhance drainage, and prevent re-accumulation of the abscess. If the abscess is packed, patients typically have to return in 2-3 days for a repeat visit to have the packing removed. The present standard of care, gauze packing, is difficult for patients to remove alone, as the packing itself becomes impregnated with pus and blood. Additionally, the packing procedure can be painful, despite the use of local anesthetics.

A newer approach advocates for the use of a silicon string, known as a PDS loop for purposes of packing and drainage. While this approach can reduce pain, and is equally effective in terms of healing time, and treatment failure, the PDS, or Vessiloop is not readily available in emergency departments and outpatient clinics, as it is a specialized sterile surgical device used in vascular procedures. Furthermore, this procedure does not facilitate irrigation of the abscess cavity, since a much smaller incision is made. Finally, the PDS loop requires a surgical knot which may come loose.

Objective:

To investigate the use of a novel silicon packing device, the Derma-Stent™. The novel device will facilitate self removal by patients, as it has a narrower profile, and, as a nonabsorbent material, will not become saturated with bodily fluids. Although it will not absorb body fluids, it is believed that the Derma-stent will achieve the objective of wound healing by maintaining the opening of the surgical incision.

Hypothesis:

The acceptability of self removal will be significantly higher for the novel device.

Study Protocol:

ED Visit

1. Abscess measured by ultrasound. Study will be performed by a trained research assistant, and will be verified by a physician certified to interpret soft tissue sonographic images.
2. Abscess photographed, with measurement tape, to allow for objective measurement of skin induration and erythema.
3. Abscess will be incised and drained, utilizing standard of care technique, with local anesthetic
4. Packing performed according to randomization group.
5. Sterile dressing applied.
6. Subject completes assessment form - pain scale.
7. Practitioner fills out assessment form - ease of use.

Follow up visit 1 - 3-5 days

1. Removal of packing. Subjects will be asked to remove packing on their own under supervision of the physician. Physician will remove the packing if they not able to.
2. Measurement of abscess diameter and volume, utilizing measuring tape, photograph, and point of care ultrasound.
3. Practitioner and subject assessment form as above, but adding ease of procedure, and likelihood that subject would have removed packing at home.

Follow up visit 2 - 24-32 days

1. Assessment of residual erythema and fluid collection by measurement, photograph, and US
2. Practitioner and subject assessment including global satisfaction, and satisfaction with cosmetic result.

Adverse Effects:

If physician is impressed that the wound is not appropriately at either f/u visit, antibiotics may be prescribed, and repacking may be performed, utilizing gauze packing strip. Use of antibiotics for abscess is controversial and most physicians prescribe these on a case by case basis. Antibiotics will be prescribed at the discretion of the physician and not related to the study protocol.

Population:

Convenience sample of adult patients presenting with uncomplicated cutaneous abscess amenable to bedside drainage to either DRH or SGH ED.

Sample size calculation:

As this is a hypothesis generating study, and the effect size is unknown, formal sample size calculation was not performed. 60 patients was chosen as the sample size.

ELIGIBILITY:
Inclusion Criteria:

1. ED patient > 18, < 90.
2. Abscess total dimensions (z+y+z) by ultrasound greater or equal to 5 cm.
3. Consent to participate in research protocol.
4. Assessment by attending physician that the abscess will require packing.

Exclusion Criteria:

1. Patients requiring admission for skin and soft tissue infection.
2. Abscess drainage requiring procedural sedation.
3. Abscesses requiring incision and drainage in the operating room.
4. Inability to comprehend consent and follow up instructions.
5. Prisoners.
6. Pregnant women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-12-15 (Estimated)

PRIMARY OUTCOMES:
Likelihood of self removal | 3-5 days
  Likelihood of self removal, as measured on a 1-10 Likert scale.

SECONDARY OUTCOMES:
Clinical Failure Rate | 32 days after baseline
  Defined by presence of: fever, increase in maximal diameter of erythema, worsening of wound swelling and tenderness.
Recurrence Rate of Abscess | 3-5 day and one month follow-up
  Recurrence rate of abscess at initial (3-5 day) and one month follow up.
Cosmetic Result | 3-5 day and one month
  Cosmetic result at both f/u visits, as measured subjectively by participants, utilizing a 1-10 Likert scale.
Pain during procedure and packing removal | baseline and 3-5 day
  Pain during procedure and packing removal, measured by a 1-10 visual acuity scale.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Brody, MD, MPH, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pallin DJ, Egan DJ, Pelletier AJ, Espinola JA, Hooper DC, Camargo CA Jr. Increased US emergency department visits for skin and soft tissue infections, and changes in antibiotic choices, during the emergence of community-associated methicillin-resistant Staphylococcus aureus. Ann Emerg Med. 2008 Mar;51(3):291-8. doi: 10.1016/j.annemergmed.2007.12.004. Epub 2008 Jan 28. PMID 18222564
- [Background] Qualls ML, Mooney MM, Camargo CA Jr, Zucconi T, Hooper DC, Pallin DJ. Emergency department visit rates for abscess versus other skin infections during the emergence of community-associated methicillin-resistant Staphylococcus aureus, 1997-2007. Clin Infect Dis. 2012 Jul;55(1):103-5. doi: 10.1093/cid/cis342. Epub 2012 Mar 28. PMID 22460965
- [Background] Singer AJ, Talan DA. Management of skin abscesses in the era of methicillin-resistant Staphylococcus aureus. N Engl J Med. 2014 Mar 13;370(11):1039-47. doi: 10.1056/NEJMra1212788. No abstract available. PMID 24620867
- [Background] Tsoraides SS, Pearl RH, Stanfill AB, Wallace LJ, Vegunta RK. Incision and loop drainage: a minimally invasive technique for subcutaneous abscess management in children. J Pediatr Surg. 2010 Mar;45(3):606-9. doi: 10.1016/j.jpedsurg.2009.06.013. PMID 20223328
- [Background] Ladd AP, Levy MS, Quilty J. Minimally invasive technique in treatment of complex, subcutaneous abscesses in children. J Pediatr Surg. 2010 Jul;45(7):1562-6. doi: 10.1016/j.jpedsurg.2010.03.025. PMID 20638546
- [Background] Gaszynski R, Punch G, Verschuer K. Loop and drain technique for subcutaneous abscess: a safe minimally invasive procedure in an adult population. ANZ J Surg. 2018 Jan;88(1-2):87-90. doi: 10.1111/ans.13709. Epub 2016 Sep 12. PMID 27621209